CLINICAL TRIAL: NCT06221943
Title: Investigation of Effectiveness of an Intensive Caregiver-involved Group- Based Naturalistic Developmental Behavioral Intervention Program for Autistic Preschoolers- A Pilot Randomized Controlled Trial
Brief Title: Effectiveness of Caregiver-involved Group-based NDBIs Intervention for Autistic Preschoolers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202310088RIND
Record Dates: First submitted 2024-01-15; First posted 2024-01-24 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism; Naturalistic Developmental Behavioral Intervention; Effectiveness
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): ASD preschoolers who receive group-based NDBIs intervention (aged 2-6y)
  Interventions: Behavioral: Group-based Naturalistic Developmental Behavioral Intervention; Behavioral: ASD Diagnosis
- active control group (Active Comparator): ASD preschoolers who receive one-on-one NDBIs intervention (aged 2-6y)
  Interventions: Behavioral: One-on-one Naturalistic Developmental Behavioral Intervention; Behavioral: ASD Diagnosis

INTERVENTIONS:
Behavioral: Group-based Naturalistic Developmental Behavioral Intervention — Naturalistic Developmental Behavioral Intervention (Utilized NDBI-Fi as the fidelity criteria of the intervention) provided in a group setting.
  Arms: experimental group
Behavioral: One-on-one Naturalistic Developmental Behavioral Intervention — Naturalistic Developmental Behavioral Intervention (Utilized NDBI-Fi as the fidelity criteria of the intervention) provided in an one-on-one setting
  Arms: active control group
Behavioral: ASD Diagnosis — Autism Diagnostic Interview-revised (ADI-R) and Autism Diagnostic Observation Scale (ADOS)

SUMMARY:
This is a study that investigate the effectiveness of NDBIs for autistic preschoolers delivered in group-settings and one-on-one settings. The outcome measures assess the improvements in autistic symptoms, social communication, play skills, group behaviors, adaptation, and parent stress.

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) is characterized by persistent social communication deficits and restricted behaviors. Global prevalence is 1-2%, with 1% in Taiwan. Social interaction obstacles and repetitive behaviors impact ASD individuals in various contexts, emphasizing the need for effective interventions. Current treatments focus on behavioral approaches, particularly Naturalistic Developmental Behavioral Interventions (NDBIs). NDBIs improve social engagement, cognitive development, and language skills. Parent-mediated intervention (PMI) enhances treatment effectiveness and reduces parenting stress. However, many NDBIs are conducted in one-on-one settings, limiting feasibility, especially in schools. Group-based interventions are beneficial and more feasible in the communities, but limited research exists. In Taiwan, early interventions, covered by National Health Insurance, lack intensity and parent involvement. The study aims to establish an intensive, parent-involved, group-based NDBIs program. The randomized controlled trial will assess its effectiveness in improving autistic symptoms, social and play skills, group behaviors, general adaptation, and reducing parenting stress.

ELIGIBILITY:
Inclusion Criteria:

* clinically diagnosed as Autism Spectrum Disorder
* aged 2-6 years old
* one of caregivers is able to participate treatment sessions.

Exclusion Criteria:

* having other major diseases.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Autism Treatment Evaluation Checklist | 10 minutes
  The Autism Treatment Evaluation Checklist (ATEC) is a tool with 77 items (likert-scaled 0-3) designed to evaluate treatment effectiveness for individuals with autism. It comprises four subscales: Speech/Language Communication, Sociability, Sensory/Cognitive Awareness, and Health/Physical Behavior. The reduced scores represented the improvement in these areas.The total score of the ATEC ranges from 0 to 180, with a higher score indicating greater severity of autism symptoms.
Mullen Early Scale Learning | 50 minutes
  A comprehensive measure of cognitive functioning for infants and preschool children from birth to 68 months, consisting of five subscales: gross motor, visual reception, fine motor, receptive language, and expressive language. The maximum raw score is 50 and will be transformed into T score based on the child's age, which can then be used to determine the percentile rank and scale age equivalent.
Individual Growth and Development Indicators | 15 minutes
  A play-based observational measure assessing communication, motor function, sociability, and problem solving in toddlers. In this study, we will use the subscale of communication (Early communication indicator) and sociability (Early social indicator). Each measure lasts for 6-minutes while key communication skills and social skills will be counted as number, the rate of key skills (per-minute) will be generated and used for analysis.
Structured Play Assessment | 30 minutes
  A semi-structured assessment used to measure children's spontaneous play acts. The two indicators are the play diversity and the play complexity. The play acts are hierarchically ordered into 16 play levels. Play diversity represents the number of types of play acts are displayed, while play complexity refers to the highest level of the child's play acts.
Preschool and Kindergarten Behavior Scale-Second Edition | 15 minutes
  It is a parent-report or teacher-report questionnaire targeting young children's behaviors in preschools, consisting of social skills scale and problem behavior scale. The social skills scale consists of 34 likert-scaled item (0-3), with a higher score indicating better social skills. The problem behavior scale consists of 42 likert-scaled item (0-3), with a higher score indicating more severe problem behaviors.
Vineland Adaptive Behavior Scales - Third Edition, Chinese Version (VABS-3) | 20 minutes
  It is a widely used and well validated measurement for assessing adaptive behaviors in individuals, rated by caregivers and teachers. It consists of 4 domains: communication, daily living skills, socialization, and motor skills. These domains encompass 11 subdomains, including receptive, expressive, written, personal, domestic, community, interpersonal relationships, play and leisure, coping skills, gross motor, and fine motor. The raw scores will be transformed to standard score ranged from 20 to 140 with a higher number representing better adaptation.
Autism Parenting Stress Index | 5 minutes
  This questionnaire is used to gauge parental stress from the perspective of parents or caregivers of young children with autism. The test items are grouped into three categories: fundamental social difficulties (item 1,2,11,12,13), challenging behavior management (item 3,4,5,6), and physical concerns (item 7,8,9,10). The total score ranges from 0 to 52, with 0 indicating not stressful, 1 indicating sometimes creates stress, 2 indicating often creates stress, 3 indicating very stressful on a daily basis, and 5 indicating so stressful sometimes we feel we can't cope.
Family Empowerment Scale | 5 minutes
  It is a 5-point caregiver-reported questionnaire consisting of 34 items, which is used to measure the family empowerment in caregiving for children with special needs. The score ranges from 34-170, with a higher score representing a high level of empowerment.

SECONDARY OUTCOMES:
Assessment of Preschool Children's Participation | 20 minutes
  It measures participation in children aged 2 to 5 years and 11 months. It captures involvement in play, skill development, active physical recreation, and social activities, providing a comprehensive view of their engagement in these crucial developmental areas. It assesses the diversity and frequency of the participated activities.
Repetitive Behavior Scale-Revised | 10 minutes
  It is a tool used to assess repetitive behaviors in individuals with autism spectrum disorder. It includes 43 items (likert-scaled 0-3) divided into six subscales: Stereotyped Behavior, Self-Injurious Behavior, Compulsive Behavior, Ritualistic Behavior, Sameness Behavior, and Restricted Interests, offering a comprehensive evaluation of repetitive behaviors.
Child Behavior Checklist | 20 minutes
  This parent-reported questionnaire is a comprehensive assessment tool for identifying behavioral and emotional problems in children. It includes 100 items (scored 0-3) covering multiple domains such as anxiety, depression, social issues, and aggressive behavior, providing a detailed profile of the child's psychological functioning. The score ranges from 0-200, with a higher score representing higher concern of behavior problems.
Autism Stigma and Knowledge Questionnaire | 10 minutes
  This questionnaire assesses public perceptions and understanding of autism. It includes 49 items measuring stigma, misconceptions, and accurate knowledge about autism spectrum disorder. Parents will indicate their agreement or disagreement with each statement. Of these items, 30 are correct statements, and 19 are incorrect statements, helping identify areas where educational interventions are needed to improve awareness and reduce stigma in the community.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital Yunlin Branch, Douliu, Taiwan